CLINICAL TRIAL: NCT00698867
Title: A Prospective, Non-controlled, Clinical Investigation of the Discovery™ Elbow System
Brief Title: A Clinical Investigation of the Discovery™ Elbow System
Status: Completed | Type: Observational
Sponsor: Biomet Orthopedics, LLC (Industry)
Responsible Party: Sponsor
Organization: Zimmer Biomet (Industry)
Other Study IDs: ORTHO.CR.EX001; NCT00515515 (obsolete NCT alias)
Record Dates: First submitted 2008-06-13; First posted 2008-06-17 (Estimated); Results first posted 2017-08-07 (Actual); Last update posted 2017-08-07 (Actual); Status verified 2017-04

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Avascular Necrosis; Humeral Fractures
Keywords: Total Elbow Arthroplasty; Total Elbow Replacement; Osteoarthritis; Elbow arthritis
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Osteonecrosis; Humeral Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Discovery™ Elbow: Discovery™ Elbow minimally constrained

SUMMARY:
The purpose of this study is to perform a five-year, multi-center prospective evaluation of the Discovery™ Elbow System for outcome and durability. Relief of pain and restoration of function will determine long-term clinical outcome while durability will be measured by the absence of revisions.

DETAILED DESCRIPTION:
Patient follow-up outcomes measured by the ASES score, radiographs and adverse events/revisions.

ELIGIBILITY:
Inclusion Criteria:

* Non-inflammatory degenerative joint disease including osteoarthritis and avascular necrosis.
* Inflammatory arthritis
* Revision where other devices or treatments have failed
* Correction of functional deformity
* Treatment of acute fractures or non-union about the elbow

Patient Selection factors to be considered include:

* Need to obtain pain relief and improve function.
* Ability and willingness to follow instructions including control of weight and activity levels.
* Patients who are able and willing to return for follow-up evaluations.
* Patients with a good nutritional state.
* Patients with full skeletal maturity.
* Patients of all races and gender.
* Patients who are able to follow care instructions.

Exclusion Criteria:

* Patients less than 18 years.
* Patients with marked bone loss which would preclude proper fixation of the prosthesis.
* Metabolic disorders, which may impair bone formation.
* Patients who are pregnant.
* Patients with an active or suspected infection in or around the elbow or distant foci of infections, which may spread to the implant site.
* Patients with a highly communicable disease or diseases that may limit follow-up (e.g. immuno-compromised conditions, hepatitis, active tuberculosis, neoplastic disease, etc.).
* Patients unwilling or unable to comply with a rehabilitation program for elbow replacement or who indicate difficulty or inability to return for follow-up visits prescribed by the study protocol.
* Patients who qualify for inclusion in the study, but refuse consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in need of relief from painful or disabling Joint Disease in need of total elbow replacment.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2002-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell Schenck, PhD, Study Director — Director, Clinical Research, Biomet Orthopedics, LLC
Locations (4):
- United States (4):
  - Florida Orthopedic Institute, Tampa, Florida
  - Indiana Hand to Shoulder Center, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Vanderbilt Hand Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Elbows
Period: Overall Study
Arm/Group | Discovery™ Elbow
Started | 118; 118 Elbows
Subjects With 1 Year Data | 68; 68 Elbows
Subjects With 2 Year Data | 55; 55 Elbows
Subjects With 3 Year Data | 35; 35 Elbows
Subjects With 4 Year Data | 34; 34 Elbows
Completed | 27; 27 Elbows
Not Completed | 91; 91 Elbows

BASELINE CHARACTERISTICS:
Population: Elbows with preoperative data
Arm/Group | Discovery™ Elbow
Number analyzed (Participants) | 118
Age, Customized [Number; unit: Elbows]
  Less than 20 | 0
  20-29 | 1
  30-39 | 7
  40-49 | 10
  50-59 | 24
  60-69 | 41
  70-79 | 22
  80-89 | 11
  90-99 | 2
Sex/Gender, Customized [Number; unit: elbows]
  Female | 90
  Male | 28
Region of Enrollment [Number; unit: elbows]
  United States | 118
Hand Dominance [Number; unit: elbows]
  Ambidextrous | 2
  Left | 5
  Right | 111
Primary Diagnosis [Number; unit: elbows]
  Functional Deformity | 1
  Humeral Fracture | 20
  Osteoarthritis | 8
  Other | 13
  Other Inflammatory Arthroses | 1
  Rheumatoid Arthritis | 52
  Traumatic Arthritis | 15
  Ulnar Fracture | 2
  Recurrent Dislocation/Stability | 5
  Revision Surgery | 1

OUTCOME MEASURES:

1. Primary Outcome: American Shoulder and Elbow Society Score (ASES) Pain Assessment
Description: This is a patient reported outcome measure that indicates the patient's pain as measured on the ASES form. The maximum pain score is 50 and the minimum score is 0. A higher pain score indicates the subject is in more pain. A lower pain score indicates less pain.
Time Frame: 5 years
Population: Discovery Elbow
Measure: Mean (Standard Deviation); unit: Scores on a scale
Units Other Than Participants: Elbows
Arm/Group | Discovery™ Elbow
Number analyzed (Participants) | 27
Number analyzed (Elbows) | 27
Scores on a scale | 5.4 (7.1)

2. Primary Outcome: Patient Derived American Shoulder and Elbow Society Score (ASES) Function
Description: This is a measure of patient function as answered by the patient. The maximum score is 36 and the minimum is 0. The maximum score represents maximum function.
Time Frame: 5 Years
Population: Discovery elbows
Measure: Mean (Standard Deviation); unit: Scores on a scale
Units Other Than Participants: Elbows
Arm/Group | Discovery™ Elbow
Number analyzed (Participants) | 27
Number analyzed (Elbows) | 27
Scores on a scale | 29.7 (7.0)

3. Primary Outcome: Patient Derived American Shoulder and Elbow Society Score (ASES) Satisfaction
Description: This is a measure of patient satisfaction as answered by the patient. The maximum score is 10 and the minimum is 0. The maximum score indicates maximum satisfaction.
Time Frame: 5 Years
Measure: Mean (Standard Deviation); unit: Scores on a scale
Units Other Than Participants: Elbows
Arm/Group | Discovery™ Elbow
Number analyzed (Participants) | 27
Number analyzed (Elbows) | 27
Scores on a scale | 8.7 (2.9)

4. Primary Outcome: Surgeon Derived American Shoulder and Elbow Society Score (ASES) Signs
Description: This is a measure of the elbow signs as reported by the investigator. Signs include various assessments of joint tenderness, impingement, and pain in range of motion. The maximum score is 39 and the minimum is 0. The maximum score indicates the most abnormal signs.
Time Frame: 5 Years
Measure: Mean (Standard Deviation); unit: Scores on a scale
Units Other Than Participants: Elbows
Arm/Group | Discovery™ Elbow
Number analyzed (Participants) | 27
Number analyzed (Elbows) | 27
Scores on a scale | 1.0 (1.8)

5. Primary Outcome: Surgeon Derived American Shoulder and Elbow Society Score (ASES) Stability
Description: Surgeon assessment of patient elbow stability. Maximum instability score is 9 and the minimum is 0. The maximum score indicates the least stability.
Time Frame: 5 Years
Measure: Mean (Standard Deviation); unit: Scores on a scale
Units Other Than Participants: Elbows
Arm/Group | Discovery™ Elbow
Number analyzed (Participants) | 27
Number analyzed (Elbows) | 27
Scores on a scale | 0.00 (0.00)

6. Primary Outcome: Surgeon Derived American Shoulder and Elbow Society Score (ASES) Strength
Description: Measure of elbow strength as defined by the investigator. Maximum score is 20 and the minimum is 0. The maximum score indicates maximum strength.
Time Frame: 5 Years
Measure: Mean (Standard Deviation); unit: Scores on a scale
Units Other Than Participants: Elbows
Arm/Group | Discovery™ Elbow
Number analyzed (Participants) | 27
Number analyzed (Elbows) | 27
Scores on a scale | 19.8 (0.8)

7. Secondary Outcome: Incidence of Surviving Elbows
Description: Proportion of elbows that did not require revision or removal
Time Frame: Up to 5 Years
Population: Subjects with complete 5 year data.
Measure: Number (95% Confidence Interval); unit: Proportion of Elbows
Units Other Than Participants: Elbows
Arm/Group | Discovery™ Elbow
Number analyzed (Participants) | 27
Number analyzed (Elbows) | 27
Proportion of Elbows | 0.9778 [0.9347 to 1.0000]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of enrollment to the time of study completion (5 year visit). The numbers at risk refer to the number of elbows implanted.
Arm/Group | Discovery™ Elbow
Serious Adverse Events (participants affected / at risk) | 17/118
Other Adverse Events (participants affected / at risk) | 32/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Discovery™ Elbow (N=118)
Left shoulder arthroplasty due to rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Infection requiring intervention (Infections and infestations) | 3 (3)
Humeral Fracture (Musculoskeletal and connective tissue disorders) | 3 (3) — Postoperative humeral fracture
Sucutaneous Abscess (Infections and infestations) | 1 (1) — Patient developed 2 subcutaneous abscesses both requiring operative intervention. One abscess was located on the right dorsal wrist and the second was located on the plantar aspect of the right foot.
Post-op Hematoma (Blood and lymphatic system disorders) | 2 (2)
GI Bleed (Gastrointestinal disorders) | 1 (1)
Loosening of total elbow (Musculoskeletal and connective tissue disorders) | 2 (2)
Non-elbow Fracture (Musculoskeletal and connective tissue disorders) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Elbow Contracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Failed Ulnar Bushing (Musculoskeletal and connective tissue disorders) | 1 (1)
Resection of Distal Ulna (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Discovery™ Elbow (N=118)
Fracture Near Operative Site (Musculoskeletal and connective tissue disorders) | 10 (10)
Patient Fell (Musculoskeletal and connective tissue disorders) | 6 (7)
Stitch Abscess (Infections and infestations) | 1 (1)
Olecranon and Triceps Deficiency (Musculoskeletal and connective tissue disorders) | 1 (1)
Motor Vehicle Accident (Musculoskeletal and connective tissue disorders) | 1 (1)
Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Elbow Bursitis (Musculoskeletal and connective tissue disorders) | 2 (2)
Perforation Anterior Medical Proximal Ulna (Musculoskeletal and connective tissue disorders) | 1 (1)
Ulnar Neuropathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Foreign Body Reaction/Excision Olecranon Mass (Musculoskeletal and connective tissue disorders) | 1 (1)
Elbow Squeaking (Musculoskeletal and connective tissue disorders) | 1 (1)
MCP Replacement (Musculoskeletal and connective tissue disorders) | 1 (1)
Coagulase Negative Staph Infection (Infections and infestations) | 1 (1)
Posterior Screw Backing Out (Musculoskeletal and connective tissue disorders) | 1 (1)
Humeral radiolucency (Musculoskeletal and connective tissue disorders) | 1 (1)
Humeral Component Loosening (Metabolism and nutrition disorders) | 1 (1)
Posterior Nerve Palsy (Musculoskeletal and connective tissue disorders) | 1 (1)
Painful Lateral Elbow (Musculoskeletal and connective tissue disorders) | 1 (1)
Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Wound Drainage (Infections and infestations) | 2 (2)
Olecranon Impingement (Musculoskeletal and connective tissue disorders) | 1 (1)
Insidious Onset Edema Elbow (Infections and infestations) | 1 (1)
Ectopic Bone Formation (Musculoskeletal and connective tissue disorders) | 1 (1)
Elbow Contracture (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A publication which uses data in addition to the authors will be reviewed by all who have contributed data, and all of the contributors will be recognized. All publications will be reviewed by BIOMET at least 30 days prior to publication.